CLINICAL TRIAL: NCT01242891
Title: A Prospective, Multi-center, Single Arm Study to Assess the Safety and Probable Benefit of the Berlin Heart EXCOR® Pediatric Ventricular Assist Device (EXCOR® Pediatric)Under a Continued Access Protocol.
Brief Title: Assess Safety and Probable Benefit of the EXCOR® Pediatric Ventricular Assist Device Under a Continued Access Protocol
Acronym: CAP
Status: Approved for marketing | Type: Expanded Access
Sponsor: Berlin Heart, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: EXCOR® Continued Access
Record Dates: First submitted 2010-11-16; First posted 2010-11-17 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Heart Failure; Cardiomyopathies
Keywords: Ventricular Assist Device; Pediatric Ventricular Assist Device
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

INTERVENTIONS:
Device: EXCOR® Pediatric Ventricular Assist Device — Extracorporeal Ventricular Assist Device
  Other Names: Berlin Heart; EXCOR®; EXCOR® Pediatric; EXCOR® Pediatric VAD

SUMMARY:
The main purpose of this protocol is to provide a mechanism for continued access for patients that would have been enrolled into the primary cohorts of the IDE study.

DETAILED DESCRIPTION:
The data collection and protocols for this study remain consistent with the main IDE study for the EXCOR® Pediatric Ventricular Assist Device. This protocol was closed at the same time as the main IDE study due to FDA approval (December 16, 2011).

ELIGIBILITY:
Inclusion Criteria:

- Severe New York Heart Association (NYHA) Functional Class IV (or Ross Functional Class IV for patients <= 6 years) heart failure refractory to optimal medical therapy, and has met at least one of the following criteria:

* INTERMACS profile status 1 or 1A, i.e. critical cardiogenic shock (low BP unresponsive to support), compromised end organ perfusion, < 24 hour survival without mechanical support; may be due to Ventricular Tachycardia (VT)/Ventricular Fibrillation (VF) (1A) OR
* INTERMACS profile status or 2A (i.e progressive decline): not in imminent danger, but worsening despite optimal inotropic therapy; may be due to VT/VF (2A) AND at least one of the following criteria: Decline in renal functions, Decline in nutritional status, Decline in mobility/ambulation

OR

* Support with extra-corporeal membrane oxygenation (ECMO) or other mechanical circulatory support device OR
* Unable to separate from cardiopulmonary bypass

  * Listed (UNOS status 1A or equivalent) for cardiac transplantation
  * Two-ventricle circulation, including cardiomypathy, repaired structural heart disease or acquired heart disease
  * Age 0 to 16 years
  * Weight >= 3 kg and <= 60 kg
  * Legal guardian (and patient if age-appropriate) understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provide written informed consent and assent prior to the procedure.

Exclusion Criteria:

* Support on ECMO for >= 10 days
* Cardiopulmonary resuscitation (CPR) duration >= 30 minutes within 48 hours of implantation
* Body weight < 3.0 kg or Body Surface Area > 1.5 m2
* Presence of mechanical aortic valve
* Unfavorable or technically-challenging cardiac anatomy including single ventricle lesions, complex heterotaxy, and restrictive cardiomyopathy
* Evidence of intrinsic hepatic disease
* Evidence of intrinsic renal disease
* Evidence of intrinsic pulmonary disease
* Hemodialysis or peritoneal dialysis (not including dialysis or continuous veno-venous hemofiltration (CVVH) for fluid removal)
* Moderate or severe aortic and/or pulmonic valve insufficiency
* Apical VSD or other compromise that is technically challenging to repair at implant
* Documented heparin induced thrombocytopenia (HIT)
* Documented coagulopathy
* Hematologic disorder
* Active Infection within 48 hours of implant (positive blood culture or White Blood Cell count >15,000 and fever > 38 degrees C)
* Documented Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
* Evidence of recent life-limiting malignant disease
* Stroke within 30 days prior to enrollment
* Psychiatric or behavioral disease
* Currently participating in another IDE or IND trial
* Patient is pregnant or nursing

Ages: 1 Day to 16 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: All Previous IDE Sites, Principal Investigator — See IDE Clinical Trials Listing for IDE Study

REFERENCES:
- See also: Berlin Heart Inc — http://www.berlinheart.com